CLINICAL TRIAL: NCT01309061
Title: Preliminary Investigation of the Effect of Human Adipose Tissue-derived Mesenchymal Stem Cell in Progressive Hemifacial Atrophy(Romberg's Disease)
Brief Title: The Effect of Human Adipose Tissue-derived MSCs in Romberg's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSC-Facial-Stem
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Progressive Hemifacial Atrophy; Romberg's Disease
MeSH Terms: conditions — Facial Hemiatrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Intramuscular infusion of Autologous Adipose Tissue derived MSCs with autologous microlipoinjection. Dose: 1x10e7 cells/500ul/lipoinjection 20ml

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of adipose tissue derived mesenchymal stem cells (MSCs) in patient with progressive hemifacial atrophy.

DETAILED DESCRIPTION:
Adipose derived mesenchymal stem cells (AdMSCs) represent an attractive and ethical cell source for stem cell therapy.

With the recent demonstration of MSC homing properties, intramuscular aplications of MSCs to cell-damaged diseases have increased.

In a human clinical trial, five patients who had suffered a progressive hemifacial atrophy( Romberg's disease) were intramuscular administered autologous hAdMSCs (1×10e7 cells/500ul) with autologous microlipoinjection one time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study.
* Age :18-75, males and females.
* Patients with symptom of hemifacial atrophy but not progress disease.

Exclusion Criteria:

* Patients with currently progressive hemifacial atrophy.
* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Subjects who don't understand purpose and method for this study.
* Patients with psychical disorder or drug and alcohol addiction.
* Participation in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in the study.
* Serious pre-existing medical conditions like Cardiovascular Diseases, Renal Diseases, Liver Diseases, Endocrine Diseases, Cancer and Diabetes Mellitus.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The volume change of fatty layer | 24 weeks
  To evaluate the volume change of fatty layer using 3D camera.

SECONDARY OUTCOMES:
Clinical lab tests | 24 weeks
  To assess the expression change of growth factors after tissue biopsy.
Fat absorption rate | 24 weeks
  To estimate the fat absorption rate using 3D computerized tomography and 3D camera.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Woo Choi, M.D.Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- ASAN Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Koh KS, Oh TS, Kim H, Chung IW, Lee KW, Lee HB, Park EJ, Jung JS, Shin IS, Ra JC, Choi JW. Clinical application of human adipose tissue-derived mesenchymal stem cells in progressive hemifacial atrophy (Parry-Romberg disease) with microfat grafting techniques using 3-dimensional computed tomography and 3-dimensional camera. Ann Plast Surg. 2012 Sep;69(3):331-7. doi: 10.1097/SAP.0b013e31826239f0. PMID 22907186